CLINICAL TRIAL: NCT02508246
Title: A Phase I Clinical Trial of AZD1775 in Combination With Neoadjuvant Weekly Docetaxel and Cisplatin Prior to Surgery in Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: WEE1 Inhibitor MK-1775, Docetaxel, and Cisplatin Before Surgery in Treating Patients With Borderline Resectable Stage III-IVB Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9168; NCI-2015-01064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9168 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-07-10; First posted 2015-07-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (WEE1 inhibitor MK-1, cisplatin, docetaxel, surgery) (Experimental): Patients receive WEE1 inhibitor MK-1775 PO BID on days 2-4, 9-11, and 16-18, and day -7 prior to course 1, day 1 for PD assessment. Patients also receive cisplatin IV on days 1 (or up to two days after last dose of WEE1 inhibitor MK-1775 lead-in is completed), 8 (or 7 days after first chemotherapy dose), and 15, and docetaxel IV on days 1, 8, and 15. Patients experiencing progressive disease undergo surgical resection. Patients not deemed surgically resectable proceed to chemoradiation as clinically indicated. Patients experiencing stable disease or partial response may receive 2 additional courses of treatment every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery; Drug: WEE1 Inhibitor AZD1775

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: WEE1 Inhibitor AZD1775 — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775

SUMMARY:
This phase I trial studies the side effects and the best dose of WEE1 inhibitor MK-1775 when given together with docetaxel and cisplatin in treating patients with stage III-IVB squamous cell carcinoma of the head and neck that may or may not be able to be removed by surgery (borderline resectable). WEE1 inhibitor MK-1775 may block the growth of tumor cells by blocking some of enzymes that are needed for tumor growth and may also help docetaxel and cisplatin work better by making tumor cells more sensitive to the drug. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving WEE1 inhibitor MK-1775 with docetaxel and cisplatin before surgery may kill more tumor cells and shrink the tumor, allowing patients to undergo surgery to remove it.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety profile and determine a maximum tolerated dose (MTD) dose of AZD1775 (WEE1 inhibitor MK-1775) in combination with weekly cisplatin and docetaxel as a neoadjuvant approach in locally advanced borderline resectable and/or surgically unresectable with high nodal burden (e.g., >= N2b disease) and judged appropriate for non-surgical definitive therapy.

II. To determine the pharmacokinetics (PK) of the combination of single doses of AZD1775 with fixed weekly dosing of docetaxel and cisplatin given on a three out of four week cycle.

III. To evaluate pharmacodynamic (PD) biomarkers of AZD1775 drug effect in head and neck squamous cell carcinoma (HNSCC) cancers, and in particular p53 mutated HNSCC patients.

SECONDARY OBJECTIVES;

I. To evaluate the preliminary activity and efficacy of the combination in terms of objective response rate in patients with borderline resectable and unresectable HNSCC and in particular, in p53 mutated HNSCC patients.

II. The rate of resectability for borderline unresectable patients will be noted post neoadjuvant therapy.

III. The rate of unresectable patients who underwent definitive therapy via chemoradiation.

IV. Progression-free survival will be noted as part of the preliminary efficacy determination of this study.

VI. During all parts of the study, patients will be monitored carefully for the development of adverse experiences and will be monitored for clinical and/or radiographic evidence of disease progression according to usual standards of clinical practice.

TERTIARY OBJECTIVES:

I. To gain mechanistic understanding of the link between p53 mutation status and disruption of immunoglobulin heavy constant gamma 2 (G2M) regulation deregulation.

II. To confirm kinase inhibition in tumor primary cultures as well as in patient tumor-derived xenografted (PDX) mice extracts, downstream signaling consequences (WEE1 G2 checkpoint kinase [WEE1]; WEE1's target, cyclin-dependent kinase 1 [CDC2]), and mechanisms of p53 synthetic lethality which sensitize cancer cells to genotoxic therapy.

OUTLINE: This is a dose-escalation study of WEE1 inhibitor MK-1775.

Patients receive WEE1 inhibitor MK-1775 orally (PO) twice daily (BID) on days 2-4, 9-11, and 16-18, and day -7 prior to course 1, day 1 for PD assessment. Patients also receive cisplatin intravenously (IV) on days 1 (or up to two days after last dose of WEE1 inhibitor MK-1775 lead-in is completed), 8 (or 7 days after first chemotherapy dose), and 15, and docetaxel IV on days 1, 8, and 15. Patients experiencing progressive disease undergo surgical resection. Patients not deemed surgically resectable proceed to chemoradiation as clinically indicated. Patients experiencing stable disease or partial response may receive 2 additional courses of treatment every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Current diagnosis of histological or cytopathological HNSCC malignancy borderline resectable stage III up to stage IVb (T1-4, N0-2, M0) or unresectable stage IV with high nodal status defined as >= N2b (by the American Joint Committee on Cancer [AJCC] 7th Edition Staging) that is amenable or appropriate for curative treatment; borderline resectability is assessed; NOTE: surgical unresectability will be defined as the combination of the treating surgeon's judgment of unresectability plus one of the following objective criteria:

  * Encasement of tumor or nodes to the carotid artery or 3/4 encasement of the carotid artery
  * Involvement of prevertebral musculature
  * Need for glossectomy or extensive glossal resection where functional outcome is considered unacceptable to surgeon or patient
  * Involvement of the cervical spine
  * Severe, unacceptable functional deficit that would result from any proposed definitive surgical resection

    * NOTE: the principal investigator (PI) of the study, Dr. Mendez, is a surgical ear, nose and throat (ENT) (head and neck) oncologist and all HNSCC cases will be discussed at the University of Washington/Seattle Cancer Care Alliance weekly tumor conference where two other ENT surgical oncologists, and co-investigators in this study, will help assess resectability; as surgical unresectability may vary from patient to patient based on individual anatomy, treating physicians may, with the approval of the surgical team, declare a tumor not meeting the above criteria to be unresectable; in this case, the reason for unresectability should be documented in the medical record; medical co-morbidity and poor performance status may not be used to declare a patient unresectable
* Patients must all have available tumor tissue for biopsy and not have any bleeding diathesis and/or chronic anticoagulation that cannot be stopped for the biopsy
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Absolute neutrophil count (ANC) > 1500/uL
* Hemoglobin > 9 g/dL
* Platelets > 100,000/uL
* Total bilirubin within 1.5 times the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times ULN
* Creatinine must be < 1.5 ULN or creatinine clearance must be > 50 mL/min (calculated by Cockcroft and Gault equation)
* International normalized ratio (INR) < 1.5 times ULN
* The expanded cohort will consist of predominantly (> 50%) p53 mutated HNSCC patients at the MTD
* Willingness to use a medically acceptable method of contraception throughout the study period and for 4 weeks after the final administration of AZD1775 or longer if needed as per chemotherapies' product information (all subjects)
* For female subjects with reproductive potential: a negative serum pregnancy test

Exclusion Criteria:

* Non-squamous cell carcinomas of the head and neck region i.e. nasopharyngeal carcinoma (World Health Organization [WHO] type II and III) and salivary gland carcinomas
* Severe uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, uncontrollable hypertension or any other condition or circumstance that could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives
* Prior treatment with any of the chemotherapy medications (cisplatin or docetaxel) for HNSCC or with AZD1775
* Prior bone marrow transplant or history of organ transplant requiring the need for any chronic immunosuppressive medications
* Prior radiation to any of the field required to treat the tumor
* Any distant metastatic disease
* Major psychiatric disorders which would limit compliance
* Neuropathy grade 2 or higher
* History of prolonged QT syndrome or electrocardiogram (ECG) at screening QT interval corrected for heart rate (QTc) of > 470 ms with Bazett's or Fridericia's formula
* Active infection requiring systemic antibiotic therapy or causing fever (temp > 100.5 degrees Fahrenheit [F] or 38.1 degrees Celsius [C]) within 1 week prior to dosing with AZD1775
* Pregnant or breast-feeding females
* Second primary malignancy within 3 years (not including in situ carcinoma of the cervix, non-melanoma skin cancer or low-grade [Gleason score =< 6] localized prostate cancer) at the time of consideration for study enrollment
* Known prior severe allergic/hypersensitivity to the chemotherapy or any of the components of the study treatment
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow and retain the formulated oral product or previous significant bowel resection that would preclude adequate absorption of AZD1775
* Inability or unwillingness to abstain from taking any medications or herbal supplements that are moderate or strong inducers of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) at least 1 week prior dosing with AZD1775 and while on study treatment
* Pre-existing hearing impairment (patients who are willing to accept risk of further impairment will be considered after audiologic testing)
* Patients taking live vaccines including yellow fever vaccinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events graded according to the NCI CTCAE version 4.03 | Up to 2 years post-treatment
  Summary tables and graphic displays, as appropriate, will be prepared to examine the distribution of these toxicities per cycle.
MTD of AZD1775, based on the incidence of dose limiting toxicity (DLT), graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 28 days
  DLT is defined as any adverse event judged by the investigator to be drug-related (i.e., causality rated as possible or greater) that is assessed as grade 3 or worse. Summary tables and graphic displays, as appropriate, will be prepared to examine the distribution of these toxicities per cycle.

SECONDARY OUTCOMES:
Objective response (complete response, partial response, stable disease or progressive disease) according to Response Evaluation Criteria In Solid Tumors | Up to 5 years post-treatment
Pharmacodynamic profile of AZD1775 | Time of surgery or up to day 29
  Pharmacodynamic parameters will be studied during lead-in monotherapy to determine target engagement, mainly phosphorylated WEE1 and CDC2. Prior to treatment normal tissue in the opposite side of the tumor in the oral mucosa will be used for controls. Biological specificity will be verified by assessing the phosphorylated state of WEE1 and downstream effector molecules: total CDC2, ptyr15 CDC2, for G2/M. Other relevant biomarkers and molecular or genetic analyses may be performed.
PK profile of WEE1 inhibitor MK-1775 with docetaxel and cisplatin | Pre-dose and at 1, 2, 4, 6, and 8-10 hours on days 2 and 4 of course 1, and pre-dose on day 3 of course 1
  Maximum concentration and mean terminal half-life will be focused on during PK analysis.
Progression-free survival (PFS) duration | Up to 5 years post-treatment
  PFS will be determined in days or weeks and waterfall plots and graphical data will be provided where suitable.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Mendez, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States